CLINICAL TRIAL: NCT02679066
Title: Short Forearm Casting Versus Below-elbow Splinting for Acute Immobilization of Distal Radius Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of consistent enrollment, follow up and results
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00087273
Record Dates: First submitted 2016-01-27; First posted 2016-02-10 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar-tong splint (Active Comparator): Patients are placed in a sugar-tong splint for immobilization of the distal radius fracture.
  Interventions: Device: Sugar-tong splint
- Short Forearm Cast (Active Comparator): Patients are placed in a short forearm cast, with bivalve, for immobilization of the distal radius fracture.
  Interventions: Device: Short forearm cast

INTERVENTIONS:
Device: Sugar-tong splint — Plaster immobilization including the elbow
  Arms: Sugar-tong splint
Device: Short forearm cast — Fiberglass immobilization with elbow free
  Arms: Short Forearm Cast

SUMMARY:
There is no consensus regarding the need to immobilize the elbow in immediate immobilization of closed distal radius fractures post-reduction. Decreased functionality of the upper extremity is a notable morbidity associated with below-elbow splinting of distal radius fractures post-reduction. Few studies have provided evidence comparing sugar tong splinting versus short-arm casting as methods of immediate post-reduction immobilization. The study will randomize patients with close distal radius fractures to short forearm casting versus sugar tong splinting with close follow up including radiographic and clinical evaluation.

This will provide guidance regarding the need for short forearm cast immobilization versus sugar tong splinting in early maintenance of reduction of closed distal radius fractures, as well as functional effects of sugar tong splinting versus short forearm casting.

DETAILED DESCRIPTION:
Objectives (include all primary and secondary objectives)

To determine the success of sugar tong splinting versus short arm casting for maintenance of reduction of closed distal radius fractures and to compare the functional outcomes in patients treated with sugar tong splinting versus short forearm casting as guidance for immediate post-reduction immobilization of these fractures.

Primary objectives:

Background (briefly describe pre-clinical and clinical data, current experience with procedures, drug or device, and any other relevant information to justify the research)

* Koval et al. randomized patients to long-arm versus short-arm splinting of post-reduction closed distal radius fractures and reported comparable maintenance of reduction with better functional scores in patients immobilized in a short-arm splint and thus recommended this method for immediate post-reduction immobilization of closed distal radius fractures (Bong et al. 2006).
* Grafstein et al. randomized 101 adult patients with closed distal radius fractures to sugar tong splinting versus above-elbow circumferential casting versus above-elbow volar-dorsal splinting for immediate post-reduction immobilization and followed patients closely for 3 to 4 weeks. They reported no significant difference in loss of reduction, pain scores, range of motion, or Activities of Daily Living (ADLs) between the three methods of immobilization and thus recommended treatment with any method with which the treating physician is most comfortable (Grafstein et al., 2010).
* Millet and Rushton randomized 99 women with closed distal radius fractures to below elbow plaster casts versus initial plaster casting followed by flexible casting to allow early joint range of motion and reported increased comfort, grip scores and joint mobility in early treatment period without negative effects of early motion and thus concluded that early mobilization can be a beneficial treatment option (Millet and Rushton, 1995).
* Pool prospectively studied range of motion and radiographic parameters over a two year period in over 200 patients with Colles' fractures treated with five different combinations of above- and below-elbow immobilization and concluded that while all patients went onto union and adequate function, those immobilized in above-elbow plaster lost some degree of supination. He found no benefit to above-elbow immobilization and recommended only below-elbow post-reduction immobilization (Pool, 1973).
* Sarmiento reviewed a case series of 44 patients with intra-articular distal radius fractures treated initially with an above-elbow cast initially and transitioned early to a brace allowing elbow and wrist range of motion while restricting pronation-supination and concluded that although fracture collapse did occur, functional results were good and the early mobilization reduced the stiffness and incapacitation associated with treatment of distal radius fractures (Sarmiento et al.)

Study Procedures

1. Study design, including the sequence and timing of study procedures (distinguish research procedures from those that are part of routine care).
2. Study duration and number of study visits required of research participants.
3. Blinding, including justification for blinding or not blinding the trial, if applicable.
4. Justification of why participants will not receive routine care or will have current therapy stopped.
5. Justification for inclusion of a placebo or non-treatment group.
6. Definition of treatment failure or participant removal criteria.
7. Description of what happens to participants receiving therapy when study ends or if a participant's participation in the study ends prematurely.

   * Prospective, randomized, controlled trial
   * One hundred twenty adult patients with closed fractures of the distal radius will be randomized to below-elbow, sugar-tong splinting versus short arm casting for immediate post-reduction immobilization.
   * Residents will undergo a teaching session specifically for instruction on sugar tong splinting versus short arm casting. On-call resident will have access to an electronic folder containing randomization of patient to sugar tong splint versus bi-valved short arm cast. All reductions will be performed under local hematoma block with 1% lidocaine and traction and less than three attempts at reduction.
   * Patients will follow up at one, two and four weeks for repeat Anteroposterior (AP) and lateral radiographs of the forearm to measure radiographic parameters to determine maintenance of reduction and will complete the Disabilities of the Arm, Shoulder and Hand Score (DASH) for functional scoring of the upper extremity at two weeks.
   * Maintenance of reduction, as defined below, will be compared between splint constructs overall and in stable versus unstable fractures in each immobilization group. Specific changes in radial height, radial inclination and volar tilt as continuous variables will also be compared, as will DASH scores measuring functionality.
   * Maintenance of reduction will be defined as: loss of reduction of < 2 mm radial height, < 5 degrees of radial inclination or < 10 degrees of volar tilt and/or < 2 mm intra-articular step off, in follow up radiographs as compared to immediate post-reduction radiographs (Bong et al., 2006).
   * Unstable fractures will be defined as, at injury: > 4 mm radial shortening, > 10 degrees dorsal tilt, radial-ulnar translation of radius > 2 mm, dorsal comminution > 50% diameter of radius, > 2mm intra-articular displacement (Bong et al., 2006; Stoffelen and Broos, 1998). Fractures meeting these criteria will undergo open reduction, internal fixation (ORIF) after reduction and at a later time. However, reduction parameters and maintenance of reduction will be evaluated and compared for both splinting techniques until ORIF.

Study Statistics

1. Primary outcome variable.
2. Secondary outcome variables.
3. Statistical plan including sample size justification and interim data analysis.
4. Early stopping rules.

Primary outcome variable: Maintenance of reduction

Secondary outcome variables: DASH scores, Radiographic parameters analyzed individually: radial height, radial inclination, volar tilt

Statistical plan including sample size: Sample size was calculated based on standard deviations for the above-noted outcomes variables reported in the literature and selected a sample size based on the largest calculated sample size. This was increased from 167 to 200 to account for expected dropout.

Early stopping rules: Less than 50% patient follow-up.

Risks

1. Medical risks, listing all procedures, their major and minor risks and expected frequency.
2. Steps taken to minimize the risks.
3. Plan for reporting unanticipated problems or study deviations.
4. Legal risks such as the risks that would be associated with breach of confidentiality.
5. Financial risks to the participants.

   * No medical risks outside of standard of care.
   * Patients will be treated with standard of care.
   * Research committee of Department of Orthopaedic Surgery follows the progress of the project.
   * No legal risks.
   * No financial risks.

Benefits

a. Description of the probable benefits for the participant and for society.

Below-elbow splinting is associated with decreased morbidity

ELIGIBILITY:
Inclusion Criteria:

* Adult > 18 years of age
* Closed fracture
* Isolated injury
* No prior injury to ipsilateral forearm
* Less than or equal to two attempts at reduction

Exclusion Criteria:

* Ipsilateral upper extremity injury
* Open injury or neurovascular compromise
* Greater than two attempts at reduction
* Presentation greater than 24 hours after injury

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hasenboehler, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarmiento A, Pratt GW, Berry NC, Sinclair WF. Colles' fractures. Functional bracing in supination. J Bone Joint Surg Am. 1975 Apr;57(3):311-7. PMID 1123382
- [Background] Bong MR, Egol KA, Leibman M, Koval KJ. A comparison of immediate postreduction splinting constructs for controlling initial displacement of fractures of the distal radius: a prospective randomized study of long-arm versus short-arm splinting. J Hand Surg Am. 2006 May-Jun;31(5):766-70. doi: 10.1016/j.jhsa.2006.01.016. PMID 16713840
- [Background] Grafstein E, Stenstrom R, Christenson J, Innes G, MacCormack R, Jackson C, Stothers K, Goetz T. A prospective randomized controlled trial comparing circumferential casting and splinting in displaced Colles fractures. CJEM. 2010 May;12(3):192-200. doi: 10.1017/s1481803500012239. PMID 20522283
- [Background] Pool C. Colles's fracture. A prospective study of treatment. J Bone Joint Surg Br. 1973 Aug;55(3):540-4. No abstract available. PMID 4125714
- [Background] Millett PJ, Rushton N. Early mobilization in the treatment of Colles' fracture: a 3 year prospective study. Injury. 1995 Dec;26(10):671-5. doi: 10.1016/0020-1383(95)00146-8. PMID 8745803

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugar-tong Splint | Short Forearm Cast
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar-tong Splint | Short Forearm Cast | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 60 | 125
  >=65 years | 35 | 40 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — information was lost. Study has been terminated | NA — information was lost. Study has been terminated | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — information was lost. Study has been terminated | NA — information was lost. Study has been terminated | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants] | NA — information was lost. Study has been terminated | NA — information was lost. Study has been terminated | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Maintenance of Reduction
Description: Radiologic parameters to include radial height, radial inclination and volar tilt will be measured from post-immobilization radiographs at presentation, one week, two weeks and four weeks. Maintenance of reduction will be defined as: loss of reduction of < 2 mm radial height, < 5 degrees of radial inclination or < 10 degrees of volar tilt and/or < 2 mm intra-articular step off, in follow up radiographs as compared to immediate post-reduction radiographs.
Time Frame: one month
Population: No data was collected to allow analysis.
Arm/Group | Sugar-tong Splint | Short Forearm Cast
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Disabilities of the Arm, Shoulder and Hand (DASH) Score - Upper Extremity Function
Description: This is a validated survey of upper extremity function that is administered at the two week follow up visit. The DASH is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability).
Time Frame: Two weeks
Population: No data was measured due to inconsistent collection of DASH score and patient follow up.
Arm/Group | Sugar-tong Splint | Short Forearm Cast
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 26 months
Arm/Group | Sugar-tong Splint | Short Forearm Cast
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT02679066/Prot_SAP_000.pdf